CLINICAL TRIAL: NCT02385357
Title: Effect of a Protein-enriched Drink on Muscle Function Recovery Following an Acute High Intensity Exercise Bout
Brief Title: Effect of a Protein-enriched Drink on Muscle Function
Acronym: SPORTEUS
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Puleva Biotech (Industry)
Collaborators: Universidad de Granada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Puleva
Record Dates: First submitted 2015-02-10; First posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Contracture
Keywords: Muscle function; Anaerobic power; Muscle damage
MeSH Terms: conditions — Contracture

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): 330 ml of commercial protein-enriched drink (2.5 g/100 ml of protein)
- Experimental (Experimental): 330 ml of protein-enriched drink (6 g/100 ml of protein)
  Interventions: Dietary Supplement: Protein-enriched drink

INTERVENTIONS:
Dietary Supplement: Protein-enriched drink — Participants will drink 330 ml of a protein-enriched drink (6 g/ml of protein) after a high intensity exercise that induce muscle damage (30 min running downhill with a slope of -10º)
  Arms: Experimental

SUMMARY:
There is no conclusive evidence about the effect of intake of protein-enriched drink after and acute high intensity exercise bout on muscle function and damage. The investigators aimed to study the effect of a protein-enriched drink on muscle function recovery following an acute high intensity exercise bout. The present counterbalanced, crossover, and double blind study will involve a total of 12 active men.

DETAILED DESCRIPTION:
Participants will run downhill (-10%) during 30 min at a intensity equivalent to 75-80% of their maximum heart rate (previously determined). After the exercise bout, participants will have either the placebo or the experimental drink. The investigators will measure muscle function and damage-related parameters right after the exercise as well as the three following days. This protocol will be repeated after a wash out period of 3 weeks, where the participants will have the other drink. The investigators will control exercise and diet three weeks before study entry, during the experimental week as the investigators as during the wash out period.

ELIGIBILITY:
Inclusion Criteria:

* Recreational triathletes with 2 years of experience
* Maximum oxygen uptake : ≥55 ml/kg/min
* Fat mass: 8-20% measured by dual energy x-ray absorptiometry
* Not participating in another study
* Not having ergogenic aids
* Not participating in a weight loss program
* Normal electrocardiogram
* Participants must be capable and willing to provide consent, understand exclusion criteria and accept the randomized group assignment

Exclusion Criteria:

* History of cardiovascular disease
* Diabetes or hypertension
* Medication for hypertension, hyperlipidemia, hyperuricemia or other illness.
* Smoking
* Other significant medical conditions that are life-threatening or that can interfere with or be aggravated by exercise.
* Unwillingness to either complete the study requirements or to be randomized into control or training group.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Isometric muscle strength | Change from pre- protein-enriched drink to 24, 48 and 72 hrs post- protein-enriched drink
  Isometric muscle strength of lower limbs at 90% angle.

SECONDARY OUTCOMES:
Muscle soreness of lower limbs self-reported by a visual anagogic scale and with an algometer score. | Change from post- protein-enriched drink to 24, 48 and 72 hrs post- protein-enriched drink
  Muscle soreness of the lower limbs will be self-reported by a visual anagogic scale and with an algometer score.
Power output assessed with the 30sec. Wingate anaerobic test | Change from post- protein-enriched drink to 24, 48 and 72 hrs post- protein-enriched drink
  Power output will be assessed with the 30sec. Wingate anaerobic test.
Creatine kinase | Change from post- protein-enriched drink to 24, 48 hrs post- protein-enriched drink
  Creatine kinase will be assessed after the protein-enriched drink to assess muscle recovery after a high intensity exercise bout
Urine Creatinine | Change from post- protein-enriched drink to 24, 48 hrs post- protein-enriched drink
  Concentration of creatinine in urine will be assessed after the protein-enriched drink to assess muscle recovery after a high intensity exercise bout
Resting metabolic rate | Change from pre- protein-enriched drink to 24, 48 and 72 hrs post- protein-enriched drink
Time limit (time that the participant is able to run 90% of his determined maximum aerobic velocity) | 24hrs after protein-enriched drink
  We will measure the time that the participant is able to run 90% of his determined maximum aerobic velocity

CONTACTS AND LOCATIONS:
Overall Officials: Federico Lara, PhD, Study Director — Puleva Biotech
Locations (1):
- Biosearch Life, Granada, Granada, Spain